CLINICAL TRIAL: NCT06752070
Title: Case Studies of Child Care and Development Fund Lead Agencies' Consumer Education Strategies
Status: Active, not recruiting | Type: Observational
Sponsor: National Opinion Research Center (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency); Urban Institute (Other)
Responsible Party: Principal Investigator, Rupa Datta, Vice president and distinguished senior fellow, National Opinion Research Center
Other Study IDs: 102241-0001-004; HHSP233201500048I-75P00120F370 (Other Grant/Funding Number: Administration for Children and Families, U.S. Department of Health and Human Services)
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Searching for and Selecting Child Care in the US
Keywords: Parent consumer education strategies; CCEE search; case studies; semi-structured interviews; focus groups

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Administration for Children & Families (ACF) has contracted with NORC at the University of Chicago (NORC) to conduct a study examining consumer education and parental choice in child care and early education (CCEE). The purpose of this study is to conduct case studies with up to six states, territories, or tribes to document innovative or promising strategies that help parents looking for and selecting CCEE that meet their family's needs. The research team identified select strategies to examine based on findings from an environmental scan the project team previously completed that was designed to uncover consumer education strategies that are innovative or promising in terms of reaching families, and go beyond federal requirements. The study team selected five states and one territory: California, Georgia, Minnesota, New Hampshire, Texas, and the Commonwealth of the Northern Mariana Islands (CNMI).

This study collected information about (a) how and why each case chose to use the identified consumer education strategy; (b) efforts involved to develop and implement the strategy; (c) barriers and facilitators to implementation; and (d) parent's perspectives on and knowledge of the resources available to them to help look for and select CCEE.

The study team designed the case studies to obtain data from people with a vested interest in or leadership role related to consumer education strategies and from parents of young children. The team designed semi-structured interviews and focus groups to be conducted via Zoom.gov with participants from each site. Example participants are CCDF administrators and staff and Child Care Resource & Referral (CCR&R) agency staff. Second, the study team designed virtual focus groups to be conducted with up to 20 parents in each selected site who had a child under the age of six and were using or had previously looked for CCEE. The team also developed a short web-based survey to administer to parents participating in focus groups to capture descriptive information about study participants, such as demographic characteristics and receipt of child care subsidies.

DETAILED DESCRIPTION:
Study aims: This study aims to identify innovative or promising consumer education strategies that states, territories, and tribes can use. This information may support peer learning and innovation to advance the field. The information is not intended to assess the effectiveness or impact of consumer education strategies, and this limitation will be clearly stated in written materials associated with the study. ACF will also use this information internally to inform future planning and decision-making.

Research questions:

What motivated the state/territory/tribe to use the identified current consumer education strategy, and how was it selected? What successes has the state/territory/tribe observed in terms of improving the timing of outreach to families, raising awareness of child care search resources and care options, and supporting families' care searches? What, if any, implementation challenges did the state/territory/tribe experience? Which types of families were hardest to reach with the strategies implemented, and why? What is involved in searching for CCEE? When, how, and why do parents search? What supports do parents need to help them search for and make decisions about care under different circumstances (e.g., first-time parent)? How aware are families of sources of child care consumer education in their state/territory/tribe, and what are their perspectives on them? What do they think would be useful to them in their search for care?

Recruitment: Within each selected site, the study team purposely selected case study participants to bring a range of perspectives to address the study's research questions regarding the state or territory's strategy. In addition, the study team recruited parents across the six selected sites using a flyer distributed with the help of site agency staff and others who participated in the case studies. The recruitment flyer included information about study eligibility, requirements for participation in the focus groups, information about the $60 thank-you gift card participants received for their time, and the research team's contact information.

Data collection methods: The study team conducted virtual semi-structured interviews and focus groups as the primary methods of data collection along with a short survey administered to participating parents. Semi-structured interviews were selected for collecting data from case study participants. This selection was done as it allows for an in-depth understanding of each participant's perspective while also permitting enough flexibility to adjust the questions depending on the specific strategy's characteristics and how it is implemented. Data collection was completed by a trained researcher via Zoom.gov.

For collecting semi-structured interviews with case study participants, the study team used three instruments. First, the team developed and used an interview guide for the CCDF state and territory administrators. This guide included questions about the background, motivation, and history of the strategy; the strategy's implementation challenges and successes; and lessons learned. Second, the team developed and used an interview guide for interviewing staff in the agency/organization(s) contracted to provide consumer education services (may be a CCR&R or other local community organization). This guide included questions about participants' background, the community context, the range of consumer education strategies, the development of the focus strategy, and implementation challenges and successes. Third, the research team developed and used semi-structured interview guides that could be tailored to multiple positions and community members. This guide included questions about participants' background, the community context, perceived need for consumer education, perspectives and roles in the design and implementation of the focus strategy.

Focus groups were used as a method of data collection to allow the team to learn about perceptions, attitudes, opinions, beliefs, and views of parents. Focus groups were completed by a trained researcher. Most focus groups were completed with several parents, but if a parent could not join a focus group time, a team member conducted a one-on-one interview with them instead. The team developed and used a focus group moderator's guide and a brief questionnaire. The semi-structured focus group guide was developed to accommodate various scenarios and included questions and probes from which the facilitator could choose based on the participants present. The focus group questions included questions about parents' child care search experiences, sources of information they used and found helpful or not as helpful and why, and their thoughts on the selected consumer education strategy.

At the end of the focus group, the study team shared a link with participants, who were directed to complete a brief web-based questionnaire designed to capture demographic information and current subsidy receipt.

Data Analysis: Each interview and focus group was audio recorded, and recordings were sent to a third-party service for a transcription. The lead senior researcher is analyzing key themes that emerge from each site to describe each site's strategy. Content from the interviews is being analyzed for each site to be integrated in site-specific documents. The team plans to develop final public documents with findings for each site organized into the following categories: background, description of case study participants, description of community context, overview of selected strategy, factors related to the success of the strategy, and lessons learned about the strategy.

The focus groups recordings are being transcribed, coded, and analyzed in NVivo software by two trained research associates. The researchers are using a combination of inductive and deductive coding that consist of developing a set of codes a priori and adding to the code scheme as new topics emerge. For this, the research team first developed a coding scheme a priori reflecting the main focus group topics and questions (e.g., sources of information used). The two researchers conducted three test coding sessions. After the first transcript was double-coded, the researchers checked the inter-rater reliability calculating kappa coefficients in NVivo for codes and subcodes and discussed points of disagreement or misalignment. Kappa coefficient values below .3 were considered low in codes or subcodes and were identified as not applied with enough consistency. Specific rules were discussed and agreed on for these instances to improve reliability. A second and third transcript were double coded until reliability across all codes was acceptable (kappa value above .4). This process resulted in revisions to the coding scheme to clarify points of confusion and include emerging topics. Final analyses will be based on the final coding schema.

ELIGIBILITY:
Inclusion Criteria:

* Case study participants required to work in agencies in charge of the consumer education strategies. Parents of children under the age of 6, residing in each selected site to have gone through a child care search experience.

Exclusion Criteria:

* Being under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case study participants required to work in agencies in charge of the consumer education strategies. Parents of children under the age of 6, residing in each selected site to have gone through a child care search experience.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Background and history of parental education strategy | May 2023-August 2025
  Semi-structured interviews provided information about the motivations of the states/territories to use their current consumer education strategy/strategies. Information about the goal (or theory of change) of this innovation. Information on the populations (e.g., universal or some subset of families) was it intending to reach.
Factors related to the success of the strategy | May 2023-August 2025
  Semi-structured interviews provided information about what successes the state/territory observed in terms of improving the timing of outreach to families, raising awareness of child care search resources and care options, and supporting families' care searches. Information on how states and territories are measuring success. Information on the key ingredients of successful implementation.
Lessons learned about the strategy | May 2023-August 2025
  Semi-structured interviews provided information about the implementation challenges that the state/territory experienced. Information on the types of families that were hardest to reach with strategies implemented and reasons behind those difficulties. Description of the challenges that remain and the supports that states/territories need to be more effective.
Parents' awareness of the consumer education strategies | May 2023-August 2025
  The parent focus groups provided information about the families' awareness of sources of child care consumer education.
Primary sources of information about child care | May 2023-August 2025
  The parent focus groups obtained information about where parents may have gotten information about child care and early education (CCEE).
What parents look for when searching for CCEE | May 2023-August 2025
  The parent focus groups provided information on the characteristics that parents look for in a provider when searching for CCEE.
Most useful sources of information when looking for CCEE | May 2023-August 2025
  Parents focus groups described the information that parents found most and least helpful. Also, parental assessment of the most helpful source of information or resources when looking for CCEE.

CONTACTS AND LOCATIONS:
Locations (1):
- The Urban Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No